CLINICAL TRIAL: NCT05858918
Title: Evaluation the Effect of Ticagrelor and Clopidogrel in Stable Coronary Syndrome A Randomized Clinical Trial
Brief Title: Ticagrelor vs. Clopidogrel in Post PCI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SUMS.MED.REC.1401.351
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Stable Chronic Angina
Keywords: Percutaneous coronary intervention; dual antiplatelet therapy; major adverse cardiovascular event; P2Y12 inhibitor; ticagrelor; clopidogrel
MeSH Terms: conditions — Angina, Stable | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Intervention Model Description: comparing two antiplatelet drugs , head to head, randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- clopidogrel (Active Comparator): patient post elective angioplasty and stenting receiving aspirin 80 mg and clopidogrel 75 mg PO daily
  Interventions: Drug: Clopidogrel
- ticagrelor (Active Comparator): patient post elective angioplasty and stenting receiving aspirin 80 mg and ticagrelor 90 mg PO twice daily
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Treatment with dual antiplatelet drug,aspirin 80 mg PO daily with clopidogrel 75 mg PO daily
  Arms: clopidogrel
Drug: Ticagrelor — Treatment with dual antiplatelet drug,aspirin 80 mg PO daily with ticagrelor 90 mg PO twice daily
  Arms: ticagrelor

SUMMARY:
Elective PCI were included in the study. Patients were randomized into two different groups. One group took ASA 80 mg once daily and clopidogrel 75 mg once a day, and the other one took ASA 80 mg once a day and ticagrelor 90 mg twice a day. After six months of close follow-up, patients were asked to give a score to their dyspnea and asked about the major advance cardiovascular events ( MACE)

DETAILED DESCRIPTION:
Clinical data of this Randomized Clinical Trial (RCT) study was gathered from patients referred to Prof. Kojuri cardiovascular clinic (Shiraz, Iran, Email: kojurij@yahoo.com , webpage: http://kojuriclinic.com/ ) from October 2022 to March 2023. The inclusion criterion was experiencing elective percutaneous coronary intervention (PCI). Patients diagnosed with hypersensitivity to either ticagrelor or clopidogrel or the ones having any other contraindications such as active pathological bleeding, were excluded from the study. Patients who consumed anticoagulants in the course of their medical therapy were also excluded.

Basic clinical information of all patients such as diabetes mellitus (diagnosed based on ADA 2018 criteria [23]), hypertension (defined as systolic blood pressure > 130 mmHg or diastolic blood > 80 mmHg based on 2017 ACC/AHA hypertension guideline [24]), dyslipidemia, anemia (defined according to 1968 Who definition [25]), asthma (diagnosed based on 2007 NAEPP criteria [26]) , chronic obstructive pulmonary disease (diagnosed according to 2020 GOLD criteria [27]), and atrial fibrillation (AF) were recorded. Furthermore, other clinical data such as body mass index (normal; 18.5 to 24.9, overweight; 25 to 29.9 and obesity; higher than 30), left ventricle ejection fracture (LVEF), and heart failure (classified based on 2001 ACC/AHA heart failure classification [28]), history of using tobacco within the past 3 months, and past drug history were also recorded. Major bleeding was defined according to the Thrombolysis in Myocardial Infarction (TIMI) criteria: intracranial bleeding, hemorrhage with a hemoglobin decrease of at least 5 g/dL, or fatal bleeding that caused death within 7 days [29].

Patients were asked to give a score to their dyspnea based on the 10 point Likert scale before undergoing PCI. Score 1-3 were considered mild, score 4-7 were considered moderate, and score 7-10 were considered severe. Patients were randomized using the Block randomization method with block size=4 into two different groups. One group took acetylsalicylic acid (ASA) 80 mg once daily and clopidogrel 75 mg that is produced by Sanofi company available in market as Plavix once a day, and the other one took ASA 80 mg once a day and ticagrelor 90 mg that is produced by Abidi company available in market as Brilavus twice a day.

The patients were completely informed about the advantages and disadvantages of the study, and inform consents were taken from participants. Patients who desired not to participate were excluded from the study. Participants were told to take their medications regularly, and they were also encouraged to call us immediately if they faced any medical problem for further investigation.

After six months of close follow-up, patients were asked to give a score to their dyspnea happened after PCI, based on the 10 point Likert scale. They were also asked about having dyspnea on exertion, paroxysmal nocturnal dyspnea (PND), any bleeding such as GI bleeding, and occurrence of major adverse cardiovascular event (MACE; defined as acute coronary syndrome (ACS), stroke, revascularization, hospitalization due to heart failure, and cardiac death.) [29] We followed the patients by using their phone numbers which were obtained at the beginning of the study.

For statistical analyses we used IBM SPSS software version 25. Independent-sample t tests and one-way ANOVA were used for parametric variables. The Mann-Whitney U test and Kruskal-Wallis test were used for nonparametric data. Values of p <0.05 were considered significant.

The study protocol was based on Helsinky declaration, all patients were filled the written consent, The study protocol was approved by Ethical committee of Shiraz University of medical sciences under the number of IR.SUMS.MED.REC.1401.351.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing elective percutaneous coronary intervention (PCI).

Exclusion Criteria:

* Patients diagnosed with hypersensitivity to either ticagrelor or clopidogrel
* Active pathological bleeding
* Patients who consumed anticoagulants in the course of their medical therapy

Ages: 50 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
dyspnoea | 6 months
  feeling discomfort with respiration, based on 10 grade Likert grade ( minimum 0 and maximum 10, higher worse)
Number of patients with major adverse cardiovascular events | 6 months
  post angioplasty and stenting patients who developed major events, acute coronary syndrome (ACS), stroke, revascularization, hospitalization due to heart failure, and cardiac death

SECONDARY OUTCOMES:
Number of patients with bleeding | 6 months
  post angioplasty patients who developed minor or major bleeding
PND | 6 months
  Number of patients post angioplasty who developed paroxysmal nocturnal dyspnoea ( (waking from sleep with sudden dyspnoea)

CONTACTS AND LOCATIONS:
Locations (1):
- Professor Kojuri Cardiology Clinic, Shiraz, Iran

IPD SHARING:
Plan to Share IPD: No
no data will be available to public

REFERENCES:
- [Derived] Mehdizadeh Parizi M, Golchin Vafa R, Ahmadi A, Heydarzade R, Sadeghi M, Khademolhossseini A, Amiri F, Khoshnood Mansorkhani S, Tavan A, Hosseini N, Montaseri M, Hosseini SA, Kojuri J. Comparison of Ticagrelor and Clopidogrel in Elective Coronary Stenting: A Double Blind Randomized Clinical Trial. J Interv Cardiol. 2023 Dec 26;2023:5544440. doi: 10.1155/2023/5544440. eCollection 2023. PMID 38170033